CLINICAL TRIAL: NCT00389753
Title: A Prospective, Randomized, Double Blinded Controlled Clinical Trial of the Aruba Aloë Formula F-BC-096 in the Treatment of Split Thickness Donor Sites After Wound Closure
Brief Title: Aruba Aloë Formula F-BC-096 in the Treatment of Split Thickness Donor Sites After Wound Closure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never started
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2006/326
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Hydration of Scars
Keywords: Scars; Hydratation; After Treatment
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Application of Aruba Aloë formula F-BC-096 or control

SUMMARY:
Comparison between use of Aruba Aloë formula F-BC-096 and control.

DETAILED DESCRIPTION:
Patients with two equal donor sites will be selected for inclusion. After wound healing one donor site will be treated with Aruba Aloë Formula F-BC-096 while a control product will be applied to the second site.

If pressure garments are applied they must be equal for both donor sites. During follow-ups objective methods will be used to evaluate elasticity and colour of the scar.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have two similar donor sites, identical in depth and wound treatment.
* Healing time of both donor sites may differ by 3 days maximum.
* Flux values determined by Laser Doppler Imaging before commencement of the therapy must be approximately similar.
* If possible, the donor sites to be compared must have the same location.
* Patient compliance with therapy in relation to the protocol is necessary. In case of pediatric patiënts this depends on collaboration of the parents.
* For the two donor sites to be compared, the entire after-treatment concerning pressure garments or eventual silicone sheets must be equal for both donor sites.
* Patients must be available for regular and necessary follow-up.
* Possibility to finish all measurements during follow-up visits.
* Written authorisation of the patient, family or parents is required.

Exclusion Criteria:

* Donor sites are not similar (not identical in: depth, wound treatment, healing time and flux values)
* Children requiring sedation for LDI of donor sites
* Not following the complete treatment schedule or missing some evaluations during the follow-up period
* Patient has any condition(s) that seriously compromises the patient's ability to complete this study.
* Patient has participated in another study utilizing an investigational drug or device within the previous 30 days
* Patient has one or more medical condition(s), diabetes, including renal, hepatic, hematologic, neurologic, or immune disease that in the opinion of the investigator would make the patient an inappropriate candidate for this study
* Patients wish to terminate the study
* No informed consent before start of the trial

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Scar assessment after 1 month

SECONDARY OUTCOMES:
Scar assessment 3, 6 and 12 months after wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Stan Monstrey, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be